CLINICAL TRIAL: NCT01558063
Title: The Antidepressant Action of Ketamine: Brain Chemistry
Brief Title: Ketamine in the Treatment of Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NYSPI 6460; 5R01MH093637-03 (NIH)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Major Depressive Disorder
Keywords: Ketamine; Major Depressive Disorder; Treatment; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Ketamine; Sodium Chloride; Saline Solution; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Ketamine Dose 1 (Active Comparator): 0.1 mg/kg, IV (in the vein) of Ketamine and MRI scan
  Interventions: Drug: Ketamine; Procedure: Magnetic Resonance Imaging (MRI)
- Ketamine Dose 2 (Active Comparator): 0.2 mg/kg, IV (in the vein) of Ketamine and MRI scan
  Interventions: Drug: Ketamine; Procedure: Magnetic Resonance Imaging (MRI)
- Ketamine Dose 3 (Active Comparator): 0.3 mg/kg, IV (in the vein) of Ketamine and MRI scan
  Interventions: Drug: Ketamine; Procedure: Magnetic Resonance Imaging (MRI)
- Ketamine Dose 4 (Active Comparator): 0.4 mg/kg, IV (in the vein) of Ketamine and MRI scan
  Interventions: Drug: Ketamine; Procedure: Magnetic Resonance Imaging (MRI)
- Ketamine Dose 5 (Active Comparator): 0.5 mg/kg, IV (in the vein) of Ketamine and MRI scan
  Interventions: Drug: Ketamine; Procedure: Magnetic Resonance Imaging (MRI)
- Saline Solution (Placebo Comparator): Saline infused over 40 minutes and MRI scan
  Interventions: Drug: Saline; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Ketamine — Single dose of 0.1, 0.2, 0.3, 0.4 or 0.5 mg/kg of ketamine given intravenously over 40 minutes.
  Other Names: Ketalar
  Arms: Ketamine Dose 1; Ketamine Dose 2; Ketamine Dose 3; Ketamine Dose 4; Ketamine Dose 5
Drug: Saline — Single infusion of saline given intravenously over 40 minutes.
  Other Names: Saline solution
  Arms: Saline Solution
Procedure: Magnetic Resonance Imaging (MRI) — 90-minute scan during the 40-minute infusion.

SUMMARY:
Depressed patients will be offered experimental treatment with a new, potentially fast-acting antidepressant called ketamine while being scanned by magnetic resonance imaging (MRI) to measure the chemical effect of the drug. Ketamine will be given in a dose of 0.0 (placebo), 0.1, 0.2, 0.3, 0.4, or 0.5 mg/kg. If a patient does not respond to ketamine after the first infusion, it may be because s/he received ketamine placebo or the dose of ketamine was too low. In that case, an optional second scan and infusion of active ketamine (0.5 mg/kg) will be offered. This second scan will occur no later than weeks after the first scan/infusion (as scheduling permits). There is no guarantee that the patient will respond to the second ketamine infusion. Patients enrolled in the study are eligible for up to 6 months treatment with their study psychiatrist after the ketamine infusion(s).

Healthy Volunteers: Healthy controls will receive an infusion of ketamine at a single dose (0.5 mg/kg). Volunteers will only receive one MRI scan and infusion.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common illness, affecting over 14 million American adults each year. MDD is a leading cause of disability worldwide, and is responsible for huge workplace and healthcare costs. The several week delay between onset of treatment and improvement in MDD symptoms with currently available treatments further increases the burden of the disorder. Shortening this delay is a major unmet challenge in the treatment of MDD. Studies report that a single intravenous low dose of a drug called ketamine can bring about substantial improvement in depression in hours, even in patients that have not improved with other antidepressant treatments. Certain aspects of ketamine's drug action are fairly well understood, but the question remains of how these properties relate to antidepressant effect. The investigator's preliminary data support the rapid antidepressant benefit from ketamine. The investigators have used a scanner to measure the effects of ketamine on two major brain chemical transmitters and found that it causes a significant increase (more than 60%) in glutamate (Glu) and gamma aminobutyric acid (GABA) levels in the front of the brain. The investigators hypothesize that this increase in Glu and GABA levels, is responsible for the antidepressant action of the medication. Knowing how ketamine works could help to develop better medications that can be used orally and used for maintenance of the improvement seen with ketamine. The objective of the proposed dose finding study is to examine the relationship between the ketamine-induced improvement of MDD and the Glu and GABA responses to ketamine and to compare the Glu and GABA responses to ketamine in MDD and healthy subjects to better understand the pathophysiology of MDD. To achieve these aims this the investigators propose a randomized, placebo-controlled, double blind study with several different doses of ketamine. The investigators will conduct MRI scans to measure Glu and GABA before and during the ketamine treatment.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patient suffering from a major depressive episode (MDE) as part of an major depressive disorder (MDD). Patients may be psychiatric medication-free or, if on psychiatric medications, not responding adequately.
* Patient scores at least 22 on the Montgomery-Åsberg Depression Rating Scale (MADRS)
* Age range 18-65 years
* Patient is off all psychotropic and other types of drugs likely to interact with glutamate for at least 14 days before starting the study with an exception of chloral hydrate or short acting benzodiazepines for distressing anxiety or insomnia
* Subject is likely to be able to tolerate a medication washout
* Female subjects of child-bearing potential must be using an acceptable method of birth control throughout the study.
* Must be enrolled in New York Psychiatric Institute (NYSPI) study #4815

Patient Exclusion Criteria:

* Lifetime history of schizophrenia,schizoaffective illness, Bipolar Disorder, or psychosis.
* First-degree relative with schizophrenia, schizoaffective disorder, or bipolar disorder if the subject is less than 33 years old
* Significant uncontrolled physical illness particularly if it may affect the brain or glutamatergic system including blood dyscrasias lymphomas, hypersplenism, endocrinopathies, renal failure or severe chronic obstructive lung disease, autonomic neuropathies and active malignancy.
* Subjects will be excluded for baseline hypertension (BP>140/90) or significant history of cardiovascular illness
* Significant ECG abnormalities
* Lacks capacity to consent
* Patients who are actively suicidal as defined by a suicidal ideation score of 4 or 5 or suicidal behavior score > 0 on the Columbia Suicide Severity Rating Scale (C-SSRS) at in-person screening interview will be excluded from participating as outpatients and may only participate as inpatients if the independent inpatient treatment team agrees with the plan to enroll the patient.
* Electroconvulsive therapy (ECT) within the last 3 months for this episode
* Pregnancy or plans to conceive during the course of study participation
* Heart pacemaker, body implant or other metal in body
* A neurological disease or prior head trauma with evidence of cognitive impairment.
* Patients who are responding satisfactorily to antidepressant medications because they will not be washed-out for purposes of this study
* Claustrophobia sufficient to preclude MRI
* Irremovable medicinal patch
* Prior ineffective trial of, or adverse effect to, ketamine
* Subjects judged unlikely to be able to tolerate a psychoactive medication washout of 14 days
* Inadequate understanding of English
* IV drug use or history of ketamine use as a recreational drug ≥ 2 times or an adverse reaction to ketamine

Control Inclusion Criteria:

* Age 18-65
* Physically healthy
* Absence of an Axis I diagnosis (specific phobia acceptable). Absence of Borderline Personality Disorder and Antisocial Personality Disorder.
* Not on any medications known to affect glutamatergic functioning
* Female subjects of child-bearing potential must be using an acceptable method of birth control throughout the study.
* Must be enrolled in NYSPI protocol #4815

Control Exclusion Criteria:

* First degree relative with MDD; first degree relative with Schizophrenia, Schizoaffective Disorder, Bipolar disorder, if the subject is less than 33 years old, and therefore still at significant risk
* Significant active physical illness particularly if it may affect the brain or glutamatergic system including blood dyscrasias lymphomas, hypersplenism, endocrinopathies, renal failure or severe chronic obstructive lung disease,autonomic neuropathies and active malignancy.
* Subjects will be excluded for baseline hypertension (BP>140/90) or significant history of cardiovascular illness.
* Significant ECG abnormalities
* Pregnancy or plans to conceive during the course of study participation
* Heart pacemaker, body implant or other metal in body
* A neurological disease or prior head trauma with evidence of cognitive impairment.
* Claustrophobia sufficient to preclude MRI
* Irremovable Medicinal patch
* Inadequate understanding of English
* Lifetime history of substance dependence,current or past substance abuse will be excluded; IV drug use or history of ketamine use as a recreational drug ≥ 2 times or an adverse reaction to ketamine will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Grunebaum, M.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strong CE, Kabbaj M. Neural Mechanisms Underlying the Rewarding and Therapeutic Effects of Ketamine as a Treatment for Alcohol Use Disorder. Front Behav Neurosci. 2020 Dec 10;14:593860. doi: 10.3389/fnbeh.2020.593860. eCollection 2020. PMID 33362485
- [Derived] Milak MS, Rashid R, Dong Z, Kegeles LS, Grunebaum MF, Ogden RT, Lin X, Mulhern ST, Suckow RF, Cooper TB, Keilp JG, Mao X, Shungu DC, Mann JJ. Assessment of Relationship of Ketamine Dose With Magnetic Resonance Spectroscopy of Glx and GABA Responses in Adults With Major Depression: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2013211. doi: 10.1001/jamanetworkopen.2020.13211. PMID 32785636

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Dose 1 | Ketamine Dose 2 | Ketamine Dose 3 | Ketamine Dose 4 | Ketamine Dose 5 | Saline Solution
Started | 5 | 6 | 8 | 5 | 9 | 5
Completed | 5 | 6 | 8 | 5 | 9 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Dose 1 | Ketamine Dose 2 | Ketamine Dose 3 | Ketamine Dose 4 | Ketamine Dose 5 | Saline Solution | Total
Number analyzed (Participants) | 5 | 6 | 8 | 5 | 9 | 5 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.3) | 37.8 (8.2) | 38.1 (7.2) | 30.6 (9.4) | 40.2 (14.5) | 46.8 (12.3) | 38.46 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 5 | 5 | 2 | 25
  Male | 1 | 1 | 4 | 0 | 4 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 4 | 5 | 8 | 4 | 7 | 4 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders 24-hours Post-ketamine Infusion
Description: The quantitative depressive symptom ratings were collected at Baseline, Day 1 (post ketamine), Day 3 using HDRS-24 (a 24-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery). The total score can range from 0 to a maximum score of 15 with a higher score indicating a worse outcome. A "responder" was defined as an individual exhibiting a reduction in the HDRS score from baseline to 24 hours (day 1) post-treatment, and all other individuals were classified as non-responders.
Time Frame: Day 1 (post ketamine)
Measure: Number; unit: participants
Arm/Group | Ketamine Dose 1 | Ketamine Dose 2 | Ketamine Dose 3 | Ketamine Dose 4 | Ketamine Dose 5 | Saline Solution
Number analyzed (Participants) | 5 | 6 | 8 | 5 | 9 | 5
participants | 3 | 1 | 3 | 2 | 2 | 0

2. Secondary Outcome: Change in Glutamate Levels
Description: The dose-response curve as it refers to ketamine inducing a dose-dependent increase in glutamate levels with 1H Magnetic Resonance Spectroscopy (MRS) will be analyzed.
Time Frame: Baseline and 120 minutes after infusion
Population: The data was not collected at 120 minutes and therefore was not analyzed for this outcome measure.
Arm/Group | Ketamine Dose 1 | Ketamine Dose 2 | Ketamine Dose 3 | Ketamine Dose 4 | Ketamine Dose 5 | Saline Solution
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in Gamma-Amino Butyric Acid (GABA) Levels
Description: The dose-response curve as it refers to ketamine inducing a dose-dependent increase in GABA levels measured with 1H Magnetic Resonance Spectroscopy (MRS) will be analyzed.
Time Frame: Baseline and 120 minutes after infusion
Population: This data was not collected and therefore was not analyzed.
Arm/Group | Ketamine Dose 1 | Ketamine Dose 2 | Ketamine Dose 3 | Ketamine Dose 4 | Ketamine Dose 5 | Saline Solution
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- All Subjects: Includes all subjects receiving either saline or ketamine. Safety data was not collected or analyzed per dose level of ketamine.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 4/38
Other Adverse Events (participants affected / at risk) | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=38)
Active Suicidal Ideation (Psychiatric disorders) | 1 (1)
Antidepressant Misuse (Product Issues) | 1 (1)
Unrelated Medical Illness (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes